CLINICAL TRIAL: NCT05458609
Title: Lemborexant Augmentation of Naltrexone for Alcohol Craving and Sleep: A Randomized, Double-Blind, Placebo- Controlled Study
Brief Title: Lemborexant Augmentation of Naltrexone for Alcohol Craving and Sleep
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Thuy Thanh Truong, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-52091
Record Dates: First submitted 2022-07-06; First posted 2022-07-14 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — lemborexant; Naltrexone; vivitrol

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to two different arms: lemborexant plus naltrexone versus placebo plus naltrexone using a computer-generated randomization scheme.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lemborexant plus Naltrexone (Active Comparator): 10 milligrams of Lemborexant will be given daily at nighttime and 50 milligrams of Naltrexone will be given daily for a total of 4 weeks
  Interventions: Drug: Lemborexant 10 mg; Drug: Naltrexone
- Placebo plus Naltrexone (Placebo Comparator): 10 milligrams of placebo will be given daily at nighttime and 50 milligrams of Naltrexone will be given daily for a total of 4 weeks
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Lemborexant 10 mg — 10 mg of Lemborexant
  Other Names: Dayvigo
  Arms: Lemborexant plus Naltrexone
Drug: Naltrexone — 50 mg of Naltrexone
  Other Names: Vivitrol; Revia

SUMMARY:
The purpose of this study to evaluate the effects of naltrexone plus lemborexant augmentation compared to naltrexone plus placebo on cue-induced and non-cued alcohol cravings in people with alcohol use disorder and insomnia. Our secondary goals are to evaluate the effects of lemborexant plus naltrexone combination on sleep quality using self-report questionnaires and actigraph data, depression, anxiety, and suicidal ideation.

DETAILED DESCRIPTION:
Alcohol is one of the most popular substances used worldwide for thousands of years. Globally, harmful alcohol use continues to be a major public health and economic burden. The World Health Organization global status report attributed harmful alcohol use to 3 million deaths in 2016.In the United States, alcohol is the most used substance by people over the age of 12, with alcohol use disorder (AUD) affecting 14.5 million people in this age group. Hazardous alcohol use is associated with emergency room visits, overdose, driving fatalities and chronic medical conditions such as liver disease, heart disease, and hypertension.

Pharmacological interventions for AUD have expanded over the past few decades, including FDA approved and off-label medications such as naltrexone that have demonstrated efficacy in reducing alcohol cravings, consumption, and likelihood of relapse. However, the significant variability in response to treatment fuels ongoing interest in novel pharmacotherapy for AUD. A common approach involves repurposing readily available medications based on our understanding of AUD pathophysiology. In this study, we focus on the orexin system, which has been implicated in behaviors such as feeding, sleep-wake cycle, motivation, and reward associated with food, sex and substances including alcohol. The brain neuropeptides orexin A and orexin B originate in the hypothalamus and project throughout the central nervous system, activating G-protein-coupled receptors orexin 1 and 2 (OX1R and OX2R). While both orexin receptors are involved in addictive behaviors, OX1R signaling has a stronger association with reward processes whereas OX2R promotes arousal. Chronic alcohol exposure may lead to neuroadaptations in the orexin system, as observed in studies showing a positive correlation between orexin levels and severity of alcohol dependence and distress during alcohol withdrawal. Moreover, multiple animal studies have demonstrated efficacy of orexin antagonists in reducing alcohol craving, self-administration, and reinstatement of alcohol use induced by cues and stress.

The orexin antagonist lemborexant is FDA approved for treatment of insomnia. Lemborexant acts on both OX1R and OX2R and has shown efficacy in sleep initiation and maintenance compared to placebo on polysomnography and patient-report. It has demonstrated long-term safety and effectiveness without physical dependence or rebound insomnia. Compared to suvorexant, another orexin antagonist, lemborexant has greater selectivity and stronger binding for orexin receptors. Suvorexant has secondary effects on the adenosine receptor and dopamine transporter whereas lemborexant only has weak binding to melatonin 1. These differences may increase risk of misuse for suvorexant more than lemborexant. In addition, Lemborexant's longer half-life (17-19h) may be advantageous for reduction of cravings during the day.

In people with AUD, insomnia is a common problem that is associated with alcohol craving and relapse. Standard treatment for AUD with naltrexone improves cravings and other AUD outcomes, but does not improve sleep. In some cases, naltrexone may have a detrimental effect on sleep. Lemborexant may be able to target both alcohol craving/urges and insomnia when added to standard treatment with naltrexone.

ELIGIBILITY:
Inclusion Criteria:

* Admission to The Menninger clinic
* Age 18-65 years
* diagnosis of alcohol use disorder using the DSM-5 criteria confirmed with SCID-5 and
* Diagnosis of insomnia using the DSM 5 criteria, confirmed with SCID-5

Exclusion Criteria:

* unstable medical conditions (e.g. liver enzymes (ALT and AST) more than 3 times normal)
* acute alcohol withdrawal
* another drug use disorder other than nicotine and cannabis
* use of either of the study medications, naltrexone or lemborexant, within the last 30 days
* Use of any opioid medication within the past 10 days
* Use of scheduled benzodiazepines and hypnotics
* Breathalyzer positive for alcohol
* Known sensitivity to naltrexone or lemborexant
* Pregnant or breastfeeding
* Diagnosis of narcolepsy. The presence of other psychiatric illnesses, use of other psychotropic medications, and stable medical conditions will not be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Cue-induced Alcohol Cravings using the Alcohol Urge Questionnaire | 4 Weeks after Randomization
  Evaluate the effects of naltrexone plus lemborexant augmentation compared to naltrexone plus placebo on cue-induced alcohol cravings in people with alcohol use disorder and insomnia.
  Alcohol Urge Questionnaire (AUQ): an 8-item self-report questionnaire of present alcohol cravings. Each item is scored on a 1 to 7 scale (Strongly Disagree = 1 and Strongly Agree = 7). Items 2 and 7 are reverse scored. A total score is computed by averaging the item scores. Higher scores reflect greater craving. Participants will be given the AUQ shortly after going through a virtual reality scenario involving alcohol at baseline, end of week 2 and end of week 4.
Non-Cued Alcohol Cravings using the Penn Alcohol Craving Scale | 4 Weeks after Randomization
  Evaluate the effects of naltrexone plus lemborexant augmentation compared to naltrexone plus placebo on non-cued alcohol cravings in people with alcohol use disorder and insomnia.
  Penn Alcohol Craving Scale (PACS): The PACS is a 5-item questionnaire that measures alcohol craving in the past week. Scores range from 0-30, with higher scores indicating stronger cravings. The PACS will be given at baseline and weekly.

SECONDARY OUTCOMES:
Sleep Quality Using the Pittsburgh sleep quality index | 4 weeks after randomization
  Pittsburgh sleep quality index (PSQI) is a 19-item self-rated questionnaire that assesses sleep quality and disturbances. Questions are rated from 0 = no difficulty to 3 = severe difficulty. The total scores range from 0 to 21 and a score >5 is considered a significant sleep disturbance.
Insomnia Severity using the Insomnia Severity Index | 4 weeks after randomization
  Insomnia Severity Index (ISI) is a 7-item questionnaire that measures insomnia severity. Scores 8 to 14 indicates subthreshold, 15 to 21 indicates moderately severe, 22 to 28 indicates severe clinical insomnia.
Daytime sleepiness using the Epworth Sleepiness Scale | 4 weeks after randomization
  Epworth Sleepiness Scale (ESS) is an 8-item questionnaire that asks the respondent to rate on a 4-point scale (0-3) their usual chances of having dozed off or fallen asleep while engaged in eight different activities. ESS scores of 11-24 represent increasing levels of excessive daytime sleepiness.
Actigraphy to measure Total Sleep Time | 4 weeks after randomization
  The ActiGraph wGT3X-BT will measure daily total sleep time (minutes)
Actigraphy to measure sleep latency | 4 weeks after randomization
  The ActiGraph wGT3X-BT will measure sleep latency (minutes)
Actigraphy to measure wake after sleep onset | 4 weeks after randomization
  The ActiGraph wGT3X-BT will measure wake after sleep onset (minutes)
Actigraphy to measure sleep efficiency | 4 weeks after randomization
  The ActiGraph wGT3X-BT will measure sleep efficiency, which is calculated by total time asleep divided by total time in bed x 100.
Anxiety Using the Generalized Anxiety Disorder scale | 4 weeks after randomization
  Generalized Anxiety Disorder scale (GAD-7): THE GAD-7 is a self-report questionnaire that measures symptoms of generalized anxiety disorder. The participant will be given the GAD-7 at screening, baseline and weekly. Using the threshold score of 10, the GAD-7 has a sensitivity of 89% and a specificity of 82% for GAD. A score of 10 or greater on the GAD-7 indicates GAD. Cut points of 5, 10, and 15 are interpreted as mild, moderate, and severe levels of anxiety, respectively.
Depression using the Patient Health Questionnaire | 4 weeks after randomization
  The Patient Health Questionnaire (PHQ-9): The PHQ-9 a self-report questionnaire that measures symptoms of depression. The participant will be given the PHQ-9 at screening, baseline and weekly. PHQ-9 score ≥10 had a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5-9, 10-14, 15-19 and 20-27 represent mild, moderate, moderately severe, and severe depression, respectively.
Suicide Risk Using the Suicide Behavior Questionnaire-Revised | 4 weeks after randomization
  Suicide Behavior Questionnaire-Revised (SBQ-R): The SBQ-R is a 4-item questionnaire that assesses suicidal thoughts and behaviors. A score of 8 or higher indicates high risk of suicide.

CONTACTS AND LOCATIONS:
Locations (1):
- The Menninger Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swift RM, Aston ER. Pharmacotherapy for alcohol use disorder: current and emerging therapies. Harv Rev Psychiatry. 2015 Mar-Apr;23(2):122-33. doi: 10.1097/HRP.0000000000000079. PMID 25747925
- [Background] Zindel LR, Kranzler HR. Pharmacotherapy of alcohol use disorders: seventy-five years of progress. J Stud Alcohol Drugs Suppl. 2014;75(17):79-88. doi: 10.15288/jsads.2014.s17.79. PMID 24565314
- [Background] Ziolkowski M, Czarnecki D, Budzynski J, Rosinska Z, Zekanowska E, Goralczyk B. Orexin in Patients with Alcohol Dependence Treated for Relapse Prevention: A Pilot Study. Alcohol Alcohol. 2016 Jul;51(4):416-21. doi: 10.1093/alcalc/agv129. Epub 2015 Nov 22. PMID 26597795
- [Background] von der Goltz C, Koopmann A, Dinter C, Richter A, Rockenbach C, Grosshans M, Nakovics H, Wiedemann K, Mann K, Winterer G, Kiefer F. Orexin and leptin are associated with nicotine craving: a link between smoking, appetite and reward. Psychoneuroendocrinology. 2010 May;35(4):570-7. doi: 10.1016/j.psyneuen.2009.09.005. Epub 2009 Oct 13. PMID 19828259
- [Background] Moorman DE. The hypocretin/orexin system as a target for excessive motivation in alcohol use disorders. Psychopharmacology (Berl). 2018 Jun;235(6):1663-1680. doi: 10.1007/s00213-018-4871-2. Epub 2018 Mar 6. PMID 29508004
- [Background] Rosenberg R, Murphy P, Zammit G, Mayleben D, Kumar D, Dhadda S, Filippov G, LoPresti A, Moline M. Comparison of Lemborexant With Placebo and Zolpidem Tartrate Extended Release for the Treatment of Older Adults With Insomnia Disorder: A Phase 3 Randomized Clinical Trial. JAMA Netw Open. 2019 Dec 2;2(12):e1918254. doi: 10.1001/jamanetworkopen.2019.18254. PMID 31880796
- [Background] Murphy P, Moline M, Mayleben D, Rosenberg R, Zammit G, Pinner K, Dhadda S, Hong Q, Giorgi L, Satlin A. Lemborexant, A Dual Orexin Receptor Antagonist (DORA) for the Treatment of Insomnia Disorder: Results From a Bayesian, Adaptive, Randomized, Double-Blind, Placebo-Controlled Study. J Clin Sleep Med. 2017 Nov 15;13(11):1289-1299. doi: 10.5664/jcsm.6800. PMID 29065953
- [Background] Yardley J, Karppa M, Inoue Y, Pinner K, Perdomo C, Ishikawa K, Filippov G, Kubota N, Moline M. Long-term effectiveness and safety of lemborexant in adults with insomnia disorder: results from a phase 3 randomized clinical trial. Sleep Med. 2021 Apr;80:333-342. doi: 10.1016/j.sleep.2021.01.048. Epub 2021 Feb 1. PMID 33636648